CLINICAL TRIAL: NCT06675214
Title: Under Whole-course of Immunotherapy, Gradient Fractionated Radiotherapy with Concurrent Chemotherapy Versus Standard Fractionated Radiotherapy with Concurrent Chemotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma Who Achieved Partial Response After Induction Chemotherapy: a Randomized, Open-label, Multicenter, Phase III Trial.
Brief Title: Under Whole-course of Immunotherapy, Gradient Fractionated RT with CCT Versus CFRT with CCT for LANPC Who Achieved PR Post Induction Chemotherapy.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.BYAFZZX.074
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma; De-escalation Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction chemotherapy plus conventional concurrent chemoradiotherapy (Active Comparator)
  Interventions: Drug: Full course of PD-1/PD-L1 blockades; Drug: Cisplatin-based induction chemotherapy; Radiation: Standard-dose IMRT; Drug: Concurrent Chemotherapy
- Induction chemotherapy plus gradient fractioned radiotherapy and concurrent chemotherapy (Experimental)
  Interventions: Drug: Full course of PD-1/PD-L1 blockades; Drug: Cisplatin-based induction chemotherapy; Radiation: Gradient Fractionated IMRT; Drug: Concurrent Chemotherapy

INTERVENTIONS:
Drug: Full course of PD-1/PD-L1 blockades — a) Camrelizumab 200mg, b) Toripalimab 240mg, or c) Adebrelimab 1200mg will be started on day 1 of induction chemotherapy and given every 3 weeks for up to 12 cycles, or until intolerable toxicity, or disease progression or withdrawal from the treatment.
Drug: Cisplatin-based induction chemotherapy — Cisplatin-based induction chemotherapy will be given every 3 weeks for 3 cycles before radiotherapy.
Radiation: Standard-dose IMRT — GTVnx/nd:69.96Gy/33Fr/2.12Gy CTV1: 60.60Gy/33Fr/1.82y CTV2: 54.12Gy/33Fr/1.64Gy
  Arms: Induction chemotherapy plus conventional concurrent chemoradiotherapy
Radiation: Gradient Fractionated IMRT — GTVresidue: 68Gy/30Fr/2.27Gy GTVmcr: 60Gy/30F/2Gy CTV1:54Gy/30F/1.8Gy CTV2: 48GY/30F/1.60Gy
  Arms: Induction chemotherapy plus gradient fractioned radiotherapy and concurrent chemotherapy
Drug: Concurrent Chemotherapy — Cisplatin 100mg/m2 every 3 weeks for 2 cycles

SUMMARY:
This prospective trial aims to enroll patients with stage III-IVA (AJCC 8th,) locoregionally advanced nasopharyngeal carcinoma (LANPC). Under the condition of full course of PD-1/PD-L1 blockades, patients who achieved radiological partial response after 3 cycles of platinum-based chemotherapy plus PD-1/PD-L1 blockades will be randomized in a 1:1 ratio to receive gradient radiotherapy (reducing the irradiation dose of PET-CT areas without metabolic abnormalities, while maintaining adequate irradiation dose of areas with metabolic abnormalities) or standard dose radiotherapy with concurrent chemotherapy. It is expected to provide a new therapeutic option for locally advanced nasopharyngeal carcinoma at moderate risk.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO type II or type III).
2. Tumor staged as III-IVA (AJCC 8th).
3. Patients who achieved partial response according to the RECIST criteria on the basis of MRI, PET-CT and endoscopic biopsy after 3 cycles of induction therapy of platinum-based chemotherapy plus immunotherapy.
4. Eastern Cooperative Oncology Group performance status ≤1.
5. Age: 18-65 years old.
6. Adequate organ function:

   Adequate marrow function: neutrocyte count≥4×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.

   Adequate liver and kidney function: Alanine Aminotransferase (ALT)/ Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 2.5×ULN.; creatinine clearance rate ≥ 60 ml/min or creatinine of no more than 1.5 times the upper normal limit.
7. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients who are evaluated as CR or SD or PD after 3 cycles of induction therapy of platinum-based chemotherapy plus PD-1/PD-L1 blockades.
2. The laboratory examination value does not meet the relevant standards within 7 days before enrollment.
3. The images of PET-CT and enhanced MRI/CT before induction chemotherapy showed necrotic foci in the center of primary tumors or regional lymph nodes.
4. The metabolic changes shown by PET-CT images after induction chemotherapy were inconsistent with the changes in the extent of tumor invasion shown by anatomical images such as enhanced MRI/CT.
5. The primary and/or cervical metastases of patients have received prior chemotherapy, immunotherapy, targeted therapy, or surgery (except diagnostic treatment).
6. Has a known history of hypersensitivity to any components of the PD-1/PD-L1 blockades formulation or other monoclonal antibodies.
7. Has a known or suspected history of autoimmune diseases, including dementia and seizures.
8. Patients with recurrence, distant metastasis and other malignant tumors.
9. Severe heart disease, lung dysfunction, heart function, lung function below grade 3 (including grade 3)
10. Patients who underwent anti-PD-1 /PD-L1 antibody or anti-CTLA-4 antibody (or any other antibody acting on T cell synergistic stimulation or checkpoint pathway) and anti-angiogenic drugs.
11. Complications requiring long-term use of immunosuppressive drugs or systemic or local use of immunosuppressive-dose corticosteroids.
12. HIV positive; HBsAg positive and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/ml); chronic hepatitis C with blood screening positive (HCV antibody positive).
13. Has a known history of allergic reactions to the drugs in the study (gemcitabine, cisplatin, docetaxel, abraxane, paclitaxel ).
14. Has a known history of active TB (bacillus tuberculosis) within 1 year; anti-TB treatment is ongoing or within 1 year prior to screening.
15. Has received a live vaccine; or a systematic glucocorticoid therapy ; or any anti-infective vaccine (e.g. influenza vaccine, varicella vaccine, etc.) ; any Chinese anti-tumor herbs within 4 weeks prior to enrollment.
16. Pregnancy or breastfeeding.
17. Other patients who were considered unsuitable by the treating physicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years
  Defined as time from randomization to locoregional or distant metastasis relapse or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Defined as the time interval from randomization to death due to any cause.
Locoregional Relapse-Free Survival (LRRFS) | 3 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Distant Metastasis-Free Survival (DMFS) | 3 years
  Defined as the time interval from randomisation to the date of first distant metastases.
The proportion of patients with treatment related acute complications | 1 year
  The proportion of patients with treatment related acute complications according to NCI-CTC5.0 criteria and RTOG criteria.
The proportion of patients with treatment related late complications | 3 years
  The proportion of patients with treatment related late complications according to NCI-CTC5.0 criteria and RTOG criteria.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | 3 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China